CLINICAL TRIAL: NCT06374979
Title: Efficacy and Safety of Ixekizumab in Patients with Refractory Guttate Psoriasis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0047
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-02

CONDITIONS: Guttate Psoriasis
MeSH Terms: conditions — Guttate Psoriasis | interventions — ixekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ixekizumab Group (Experimental): Participants will receive an initial dose of 160 mg (two injections of 80 mg) Ixekizumab subcutaneously at week 0, followed by 80 mg at weeks 2, 4, 6, 8, 10, and 12.
  Interventions: Biological: Ixekizumab

INTERVENTIONS:
Biological: Ixekizumab — Participants will receive an initial dose of 160 mg (two injections of 80 mg) ixekizumab subcutaneously at week 0, followed by 80 mg at weeks 2, 4, 6, 8, 10, and 12.

SUMMARY:
The goal of this clinical trial is to analyse efficacy and safety of ixekizumab in participants with refractory guttate psoriasis. The main question it aims to answer is:

What percentage of participants achieved more than 90% reduction from baseline in Psoriasis Area Index （PASI 90） after 12 weeks of ixekizumab treatment? Participants will receive a 12-week treatment of ixekizumab, with follow-up visits every 2 weeks during the treatment period. Keep a diary of their symptoms and Psoriasis Area Index.

DETAILED DESCRIPTION:
This study was a single-arm, open-label, single-center multi-dose trial. Approximately 50 participants are scheduled to receive subcutaneous injection of ixekizumab for 12 weeks, with follow-up every 2 weeks during the treatment period. After the treatment period, the primary endpoint was assessed at week 16, and patients who achieved PASI 90 response were followed up at week 34 and week 52 to the medical center to assess disease recurrence or progression. To evaluate the efficacy of ixekizumab in the treatment of refractory guttate psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study and sign an informed consent form;
2. Age between 18 and 70 years, both genders are eligible;
3. Clinically diagnosed with guttate psoriasis;
4. Previously treated with traditional therapies for plaque psoriasis for more than 4 weeks (including antibiotics, topical corticosteroids, topical calcipotriene, phototherapy);
5. Current PASI score ≥ 3 or DLQI score ≥ 6;
6. Investigator assesses participants's suitability for treatment with ixekizumab;
7. No prior use of biologic agents for treatment;
8. Basic understanding of the purpose of the trial, its effects, and potential adverse events, and willing to sign the informed consent form according to the principles of the Helsinki Declaration;
9. Agree to receive regular treatment, follow-up, and undergo relevant examinations according to the clinical research protocol.

Exclusion Criteria:

1. Presence of other psoriasis phenotypes such as plaque, pustular, erythrodermic, or psoriatic arthritis;
2. Concomitant severe skin diseases, tumors, other systemic diseases (such as inflammatory bowel disease), or mental disorders;
3. Concurrent infections such as tuberculosis, HIV, hepatitis B, hepatitis C, etc.;
4. Allergy to ixekizumab;
5. Received systemic corticosteroids or immunosuppressive/immunomodulatory drugs for psoriasis treatment within the previous 4 weeks (including but not limited to methotrexate, cyclosporine, acitretin, azathioprine, hydroxychloroquine, apremilast, JAK inhibitors, etc.);
6. Participation in another clinical trial within the past 3 months;
7. Pregnant, lactating women, or those planning to become pregnant during the trial;
8. Other circumstances deemed inappropriate for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
PASI 90 response | Week 16
  The proportion of participants achieving more than 90% reduction from baseline in Psoriasis Area Index (PASI 90) after 12 weeks of ixekizumab treatment.

SECONDARY OUTCOMES:
PGA 0/1 response | Week 16
  The proportion of participants with PGA score 0 or 1 after 12 weeks of treatment.
PASI 100 response | Week 16
  The proportion of participants achieving PASI 100 after 12 weeks of treatment.
Relapse | Week 52
  Among the participants who reached PASI 90 after 12 weeks of treatment, the proportion of participants who relapsed within 52 weeks after withdrawal.

IPD SHARING:
Plan to Share IPD: No